CLINICAL TRIAL: NCT03287518
Title: Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Benefit and Tolerability of WAK2017 on Endothelial Function, Blood Pressure and Lipid Profile
Brief Title: Evaluation of the Benefit and Tolerability of WAK2017 on Endothelial Function, Blood Pressure and Lipid Profile
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Analyze & Realize (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WOA/002017
Record Dates: First submitted 2017-09-08; First posted 2017-09-19 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-10

CONDITIONS: Endothelial Function; Blood Pressure; Lipid Metabolism
Keywords: Endothelial function; Blood pressure; Lipid metabolism; EndoPAT score RHI

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel-group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Active Comparator): WAK2017 One (1) ml IP should be taken with breakfast and one (1) ml with supper every day.
  Interventions: Dietary Supplement: WAK2017
- Placebo (Placebo Comparator): The placebo liquid is identical in colour and flavor to the verum. In order to maintain the blind with respect to the odour, the placebo will contain 3% Concentrated Aged Garlic Extract (DER 0.9-1.2:1), which is considered as inactive with respect to a potential beneficial effect.
  One (1) ml IP should be taken with breakfast and one (1) ml with supper every day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: WAK2017 — WAK2017 is a solution with following active ingredients: Aged Garlic Extract. One (1) ml IP should be taken with breakfast and one (1) ml with supper every day
  Arms: Verum
Dietary Supplement: Placebo — One (1) ml IP should be taken with breakfast and one (1) ml with supper every day
  Other Names: Placebo for WAK2017
  Arms: Placebo

SUMMARY:
The main objective of the study is to evaluate the endothelial function of WAK2017. In addition the effects on the blood pressure and the parameters of lipid metabolism will be explored.

DETAILED DESCRIPTION:
The main objective of the study is to evaluate the endothelial function of WAK2017. In addition the effects on the blood pressure and the parameters of lipid metabolism will be explored.

Primary endpoint is defined as the difference in change in EndoPAT score RHI pre-dose and after 12 weeks of IP intake (visit V4 vs. V2) in comparison between the verum and placebo.

To characterize the benefit of the IP the following secondary endpoints will be analysed in comparison be-tween the verum and placebo:

* EndoPAT AI at V4 vs. V2
* SBP at V3, V4 vs. V2, respectively
* DBP at V3, V4 vs. V2, respectively
* Fasting LDL-C concentrations and non-HDL-C at V3, V4 vs. V2, respectively
* Fasting TC concentrations at V3, V4 vs. V2, respec-tively
* Fasting HDL-C concentrations at V3, V4 vs. V2, respectively
* Fasting TG concentrations at V3, V4 vs. V2, respectively
* Fasting LDL-C/HDL-C and TC/HDL-C ratio at V3, V4 vs. V2, respectively
* SCORE value at V3, V4 vs. V2, respectively
* Global evaluation of benefit by the subjects/ investigator at V4

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, 40-75 years
2. BMI 25-34.9 kg/m2
3. High normal or hypertension grade 1 blood pressure levels (130-159 / 85-99 mmHg) both at screening (mean of the 2nd and 3rd measurement during the assessment in triplicate at V1) and at baseline (mean of the 2nd and 3rd measurement during the assessment in triplicate at V2)
4. EndoPAT score (RHI): < 2.2 at V1
5. Readiness to comply with study procedures, in particular:

   * Consumption of the IP as instructed during the treatment period
   * Adhering to former diet (except consumption of max. 2 garlic cloves per week) and physical activity
   * Requirements for blood pressure / EndoPAT measurements
   * Accepting blood draws
6. Non-smoker / smoking cessation of last ≥12 months prior to V1
7. Stable body weight in the last 3 months prior to V1 (<3 kg self-reported change)
8. If allowed concomitant medications are taken this must have been stable at least during the last month prior to V1
9. Women of childbearing potential:

   * Negative pregnancy testing (beta HCG-test in urine) at V1
   * Commitment to use reliable contraception methods during the study Participation is based upon written informed consent by the participant following written and oral information by the investigator regarding nature, purpose, consequences and possible risks of the clinical study.

Exclusion Criteria:

1. Known allergy or hypersensitivity to the components of the investigational product
2. Known genetic hyperlipidemia
3. Known secondary hypertension
4. Known white-coat hypertension
5. Known type-1-diabetes
6. Uncontrolled or within the last 6 months prior to V1 diagnosed type-2-diabetes
7. Untreated or non-stabilized thyroid disorder
8. History and/or presence of clinically significant cardiovascular disease as per investigator's judgement:

   * Known congenital heart defects
   * Myocardial infarction, heart failure, angina pectoris, life-threatening arrhythmia or stroke within the last 6 months prior to V1
   * Existing thrombosis or disposition to thrombosis
9. Any other known significant or serious condition / disease that renders subjects ineligible, e.g.:

   * History of malignancy within the past 5 years prior to V1
   * Bleeding disorder and/or need for anticoagulants
   * Current psychiatric care and/or use of neuroleptics
   * Bariatric surgery in the last 12 months prior to V1
10. Any known metabolic disease, gastrointestinal disorder or other clinically significant disease/disorder which in the investigator's opinion could interfere with the results of the study or the safety of the subject
11. Known arm lymphedema (e.g. due to mastectomy)
12. Other deviation of laboratory parameter(s) at V1 that is:

    * clinically significant or
    * 2x ULN (upper limit of normal), unless the deviation is justified by a previously known not clinically relevant condition, e.g. Gilbert's syndrome)
13. Dietary habits that may interfere with the study objectives:

    * Eating disorder
    * Subjects with dietary restriction that may affect the study outcome
    * Participation in a weight loss program
14. Use of following medication/supplementation within the last 4 weeks prior to V1 and during the study, according to investigator's jugdement:

    * Drugs or supplements that can influence SBP or DBP (e.g. ACE inhibitors, diuretics, calcium channel or ß-blockers, grape seed extract, coenzyme Q10 etc.)
    * Lipid lowering drugs (affecting lipid metabolism, platelet function or antioxidant status, etc.) or dietary or health supplements (e.g. omega-3 fatty acids, green tea extract, calcium, red yeast rice, phytosterols (incl. enriched products such as e.g. Becel), oat fiber, niacin, soy protein, psyllium seed husk, glucomannan, chitosan or probiotics/prebiotics)
    * Drugs that can significantly influence cholesterol levels (e.g. corticosteroids, amiodarone, anabolic steroids)
    * Medications (e.g. statins, renin angiotensin system inhibitors, nebivolol, carvedilol, calcium channel blockers) or supplements (e.g. cocoa) that can influence vascular endothelial function and/or blood flow within the last 4 weeks prior to V1 and during the study
    * Antiplatelet agents and / or anticoagulants (e.g. warfarin, acetylsalicylic acid)
15. Use of weight loss treatment
16. Drug abuse
17. Alcohol abuse (men: ≥21 units/week, women: ≥14 units/ week; 1 unit equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits)
18. Reported participation in night shift work 2 weeks prior to V1 and/or during the study
19. Women of child-bearing potential: pregnant or breast-feeding
20. Participation in another study or blood donation during the last 30 days prior to V1
21. Any other reason deemed suitable for exclusion as per investigator's judgment

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-07-28 (Actual); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-09-15 (Estimated)

PRIMARY OUTCOMES:
Endo-PAT RHI value | Visit 2 and Visit 4 after 84 days ± 6 days after Visit 2
  Change of EndoPAT score RHI measurement Visit 2 to Visit 4. EndoPAT parameter (Reactive Hyperemia Index (RHI) will be assessed per Endo-PAT 2000 according to standardized procedures provided by the manufacturer (Itamar Medical Ltd., Israel), at Visit 2 and Visit 4

SECONDARY OUTCOMES:
EndoPAT Augmentation Index (AI) | Visit 2 and Visit 4 after 84 days ± 6 days after Visit 2
  Change of EndoPAT parameter Augmentation Index (AI) will be assessed per Endo-PAT 2000 according to standardized procedures provided by the manufacturer (Itamar Medical Ltd., Israel), at Visit 2 and Visit 4
Systolic Blood Pressure | 42 days ± 3
  Change in Systolic Blood Pressure after 6 weeks ± 3 Visit 2 versus Visit 3
Diastolic Blood Pressure | 42 days ± 3
  Change in Diastolic Blood Pressure after 6 weeks ± 3 Visit 2 versus Visit 3
Systolic Blood Pressure | 84 weeks ± 6
  Change in Systolic Blood Pressure after 12 weeks ± 6 Visit 2 versus Visit 4
Diastolic Blood Pressure | 84 days ± 6
  Change in Diastolic Blood Pressure after 12 weeks ± 6 Visit 2 versus Visit 4
Low Density Lipoprotein cholestorol (LDL-C) | 42 days ± 3
  Change in LDL-C concentration after 6 weeks ± 3 Visit 2 versus Visit 3. Blood samples will be obtained for the assessment of serum LDL-C concentrations.
Low Density Lipoprotein cholestorol (LDL-C) | 84 days ± 6
  Change in LDL-C concentration after 12 weeks ± 6 Visit 2 versus Visit 4. Blood samples will be obtained for the assessment of serum LDL-C concentrations.
non-High Density Lipoprotein cholestorol (non-HDL-C) | 42 days ± 3
  Change in non-HDL-C concentration after 6 weeks ± 3 Visit 2 versus Visit 3. Blood samples will be obtained for the assessment of serum non-HDL-C concentrations. The non-HDL cholesterol values are obtained by subtracting the HDL cholesterol value from the total cholesterol.
non-High Density Lipoprotein cholestorol (non-HDL-C) | 84 days ± 6
  Change in non-HDL-C concentration after 12 weeks ± 6 Visit 2 versus Visit 4. Blood samples will be obtained for the assessment of serum non-HDL-C concentrations. The non-HDL cholesterol values are obtained by subtracting the HDL cholesterol value from the total cholesterol
Total Cholestorol (TC) | 42 days ± 3
  Change in TC concentration after 6 weeks ± 3 Visit 2 versus Visit 3. Blood samples will be obtained for the assessment of serum Total Cholestorol (TC) concentrations.
Total Cholestorol (TC) | 84 days ± 6
  Change in TC concentration after 12 weeks ± 6 Visit 2 versus Visit 4. Blood samples will be obtained for the assessment of serum Total Cholestorol (TC) concentrations.
High Density Lipoprotein cholestorol (HDL-C) | 42 days ± 3
  Change in HDL-C concentration after 6 weeks ± 3 Visit 2 versus Visit 3. Blood samples will be obtained for the assessment of serum HDL-C concentrations.
High Density Lipoprotein cholestorol (HDL-C) | 84 days ± 6
  Change in HDL-C concentration after 12 weeks ± 6 Visit 2 versus Visit 4. Blood samples will be obtained for the assessment of serum HDL-C concentrations.
Triglycerides (TG) | 42 days ± 3
  Change in TG concentration after 6 weeks ± 3 Visit 2 versus Visit 3. Blood samples will be obtained for the assessment of serum TG concentrations.
Triglycerides (TG) | 84 days ± 6
  Change in TG concentration after 12 weeks ± 6 Visit 2 versus Visit 4. Blood samples will be obtained for the assessment of serum TG concentrations.
LDL-C/HDL-C ratio | 42 days ± 3
  Change in LDL-C/HDL-C ratio after 6 weeks ± 3 Visit 2 versus Visit 3.
LDL-C/HDL-C ratio | 84 days ± 6
  Change in LDL-C/HDL-C ratio after 12 weeks ± 6 Visit 2 versus Visit 4.
TC/HDL-C ratio | 42 days ± 3
  Change in TC/HDL-C ratio after 6 weeks ± 3 Visit 2 versus Visit 3.
TC/HDL-C ratio | 84 days ± 6
  Change in TC/HDL-C ratio after 12 weeks ± 6 Visit 2 versus Visit 4.
SCORE Value | 42 days ± 3
  The SCORE value will be assessed on V2 - V4 using the European Low Risk Chart by the European Society of Cardiology (Perk et al., 2012), during biometric assess-ment.
SCORE Value | 84 days ± 6
  The SCORE value will be assessed on V2 - V4 using the European Low Risk Chart by the European Society of Cardiology (Perk et al., 2012), during biometric assess-ment.
Global Evaluation of benefit | 84 days ± 6
  Both the subjects and investigator(s) will evaluate independently the benefit of the IP by means of a global scaled evaluation with "very good", "good", "moderate" and "poor".

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Uebelhack, MD, Principal Investigator — analyze & realize GmbH
Locations (2):
- Germany (2):
  - BioTeSys GmbH, Esslingen am Neckar, Baden Würtemberg
  - analyze & realize GmbH, Berlin

REFERENCES:
- See also: Homepage for study site in Berlin — https://proband-in-berlin.de/